CLINICAL TRIAL: NCT05242744
Title: Evaluating in Vivo PARP-1 Expression With 18F-FluorThanatrace Positron Emission Tomography (PET/CT) in Patients With Metastatic Prostate Cancer
Brief Title: FTT PET/CT in Metastatic Prostate Cancer
Status: Recruiting | Type: Observational
Sponsor: Abramson Cancer Center at Penn Medicine (Other)
Responsible Party: Sponsor
Other Study IDs: UPCC 08821; 849671 (Other: Abramson Cancer Center)
Record Dates: First submitted 2022-02-08; First posted 2022-02-16 (Actual); Last update posted 2025-07-11 (Actual); Status verified 2025-07

CONDITIONS: Prostate Cancer Metastatic
Keywords: PET/CT; PARP inhibitor

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Collected clinical or research pathology samples from primary or metastatic biopsy of prostate cancer. Research blood samples for future testing.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Metastatic prostate cancer: Men at least 18 years of age with metastatic prostate cancer may be eligible for this study .Volunteers that meet the eligibility criteria will be considered for study participation regardless of race or ethnic background. Only individuals who can understand and give informed consent will be eligible to participate in this study.
  Interventions: Drug: [18F]FluorThanatrace

INTERVENTIONS:
Drug: [18F]FluorThanatrace — Investigational radiopharmaceutical used with Positron Emission Tomography (PET/CT) imaging that may provide a non-invasive measurement of PARP-1 expression
  Other Names: [18F]FTT

SUMMARY:
Up to 30 men with metastatic prostate cancer will undergo up to 2 FTT PET/CT scans to look at PARP activity in sites of known cancer. Subjects will undergo a baseline scan prior to starting new therapy and a second, optional, post-therapy scan 1-21 days after the start of treatment. Tissue from a clinical or research biopsy will be compared to imaging measures, if available.

DETAILED DESCRIPTION:
Up to 30 evaluable patients with a histological diagnosis of prostate cancer with clinical evidence of metastatic disease who are being considered for new therapy or for a change in therapy with a PARP inhibitor, androgen deprivation therapy, and/or chemotherapy as part of their clinical care will be enrolled in this study. A pre-treatment 18F-FluorThanatrace ([18F]FTT) positron emission tomography/ computed tomography (PET/CT) scan will be done prior to the start of a new therapy regimen. PET/CT imaging will be used to evaluate PARP-1 expression in sites of prostate cancer using the investigational radiotracer [18F]FTT. This is an observational study in that [18F]FTT PET/CT will not be used to direct treatment decisions. While patients and referring physicians will not be blinded to the [18F]FTT PET/CT results, treatment decisions will be made by the treating physicians based upon clinical criteria. After injection of [18F]FTT patients will undergo a skull base to mid-thigh scan, starting at approximately 60 minutes post injection. PET/CT imaging sessions will include an injection of 12 mCi of [18F]FTT intravenously (approximate range for most studies is anticipated to be 8-12 mCi ). of [18F] FTT. Data will be collected to evaluate uptake of [18F]FTT in sites of prostate cancer, which will be compared with PARP-1 expression in tissue, when available. All evaluable patients may start new therapy following the [18F]FTT PET/CT scan. It is expected that due to patient preference and time considerations, approximately 80% will also undergo a second (optional) scan that will be performed approximately 1-21 days after new therapy has started. The second scan is obtained to evaluate whether the initiation of a PARP inhibitor and/or androgen deprivation therapy and/or chemotherapy alters [18F] FTT uptake.

ELIGIBILITY:
Inclusion Criteria:

1. Participants will be ≥ 18 years of age
2. Histologically proven prostate carcinoma
3. Clinical evidence of metastatic disease with at least one lesion identified on standard of care imaging (CT, MRI, Bone Scan, FDG or other PET/CT, Ultrasound)
4. Considered a candidate for new therapy or change in therapy with PARP inhibitor therapy and/or androgen deprivation therapy (ADT) and/or chemotherapy with or without additional agents, either on a clinical trial or as part of clinical care.
5. Participants must be informed of the investigational nature of this study and be willing to provide written informed consent and participate in this study in accordance with institutional and federal guidelines prior to study-specific procedures.

Exclusion Criteria:

1. Inability to tolerate imaging procedures in the opinion of an investigator or treating physician
2. Any current medical condition, illness, or disorder as assessed by medical record review and/or self-reported that is considered by a physician investigator to be a condition that could compromise participant safety or successful participation in the study

Min Age: 18 Years | Sex: Male
Age Groups: Adult, Older Adult
Study Population: Patients with a histological diagnosis of prostate cancer with clinical evidence of metastatic disease who are being considered for new therapy or for a change in therapy with a PARP inhibitor, androgen deprivation therapy, and/or chemotherapy as part of their clinical care.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2023-03-01 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Measurement of effect size | 21 days
  To establish effect size of change in FTT uptake before and after systemic therapy in men with prostate cancer metastasis using [18F]FluorThanatrace ([18F]FTT)

SECONDARY OUTCOMES:
Evaluation of PARP expression | 21 days
  Evaluation of PARP-1 expression in prostate cancer using measures of uptake of [18F]FTT before and after PARPi and/or androgen deprivation therapy and/or chemotherapy
Correlation with PARP-1 IHC | 6 months
  Correlation of [18F]FTT uptake measures with PARP-1 IHC expression in the tissue specimen, when available
Correlation with PARP-1 autoradiography | 6 months
  Correlation of [18F]FTT uptake measures with PARP-1 [125I]KX1 autoradiography expression in the tissue specimen, when available
Predication of clinical response | 1 year
  Determination of whether baseline and/or pre-/post-treatment changes in [18F]FTT uptake predict clinical response as measured by progression-free survival (PFS) and anatomic criteria on standard of care imaging

CONTACTS AND LOCATIONS:
Overall Officials: Neil Taunk, MD, Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania Hospital, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No